CLINICAL TRIAL: NCT06681610
Title: Modulation of the Motor Pathway by Transcranial Pulse Stimulation in People With ALS: a Pilot Randomized Trial
Brief Title: Testing Pulse Stimulation to Improve Motor Function in People With ALS: A Pilot Study
Acronym: TPS4ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-TPS-ALS-01; FUSF-RAP-S-23-00096 (Other Grant/Funding Number: Focused Ultrasound Foundation and ALS Foundation. USA)
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Transcranial Pulse Stimulation (TPS); Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: randomised, double blind, sham controlled clinical study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPS (Experimental): The stimulation will be 20 min duration as indicated in the CE mark approval. Each session involves 6,000 pulses in the hand region of the motor cortex with 3,000 on each side of the brain. The system uses a low energy flux density maximum of 0.25 mJ/mm2 accordingly with EMA and FDA guidelines (high energy is defined as > 0.5 mJ/mm2). The standard therapy involves 6 sessions in 2 weeks as indicated in the CE mark.
  Interventions: Device: Transcranial Pulse Stimulation
- sham (Sham Comparator): The transcranial pulse stimulation with the same device and the same protocol uses a membrane on the device that blocks the sound waves. Participants' motor cortex is not stimulated.
  Interventions: Device: Transcranial Pulse Stimulation

INTERVENTIONS:
Device: Transcranial Pulse Stimulation — low intensity shock-waves stimulation of the motor cortex, bilateral

SUMMARY:
The goal of this clinical trial is to assess the efficacy of TPS of the motor cortex on biomarkers and clinical endpoints in patients with ALS. The main questions it aims to answer are:

* Stage 1: Is there a change in the short intracortical inhibition (SICI) of the motor cortex from baseline to week 8?
* Stage 2: Is there a change from baseline to month 6 in the ALS functional rating scale-revised (ALSFRS-R) total score?

In stage 2, researchers will compare the group receiving the stimulation vs the group receiving a sham stimulation to see if there is a difference in motor cortex activity and in the ALSFRS-R score

Participants will receive either:

* the TPS treatment
* a sham TPS treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of sporadic ALS (definite or clinically probable) as defined by the World Federation of Neurology revised El Escorial criteria
* SVC of 50% or greater of estimated measure and presence of measurable motor evoked potential
* 21 to 80 years old and male or female

Exclusion Criteria:

* patients with fALS (based on medical history) that are unable to tolerate TMS and MRI studies or have a contraindication as described below

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the short intracortical inhibition (SICI) of the motor cortex from baseline to week 8. | baseline to week 8
Change from baseline to month 6 in the ALS functional rating scale-revised (ALSFRS-R) total score | baseline to week 24
  The ALS Functional Rating Scale-Revised Each function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0.
  Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change plasma neurofilament light chain (NfL) levels | baseline to week 4 and 8
Changes in muscle strength, assessed by the Medical Research Council (MRC) sum score | baseline to week 4 and 8
Changes in hand-held dynamometry | baseline to week 8
Differences (treated vs sham) and change in the slow vital capacity (SVC) | from baseline to month 6
Differences (treated vs sham) and change in plasma NfL levels | baseline to month 6
  Candidate biomarkers are: SOD1, Ataxin 2, C90rf72, UNC13A, TDP43, stathmin 2, NfL and NfH levels
Change in Motor Evoked Potential (MEP) Amplitudes | baseline to week 4 and 8
  ppTMS will be used to assess changes in motor cortex excitability via MEP amplitude (measured in millivolts)
Change in Resting Motor Threshold | baseline to week 4 and 8
  RMT will be recorded to assess baseline motor cortex excitability (measured as a percentage of maximum stimulator output)
Change in Intra-Cortical Facilitation | baseline to week 4 and 8
  ICF will be measured to assess synaptic excitability

OTHER OUTCOMES:
Change in biomarker SOD1 Levels in nEVs from Plasma | baseline to week 4 and 8
Change in biomarker Ataxin 2 Levels in nEVs from Plasma | baseline to week 4 and 8
Change in biomarker C9orf72 Levels in nEVs from Plasma | baseline to week 4 and 8
Change in biomarker UNC13A Levels in nEVs from Plasma | baseline to week 4 and 8
Change in biomarker TDP43 Levels in nEVs from Plasma | baseline to week 4 and 8
Change in biomarker Stathmin 2 Levels in nEVs from Plasma | baseline to week 4 and 8
Change in NfH Levels in nEVs from Plasma | baseline to week 4 and 8

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
we will provide access to protocol, SAP and ICF
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: protocol will be published as supplementary material. SAP and ICF will be provided upon reasonable request

REFERENCES:
- [Background] Voroslakos M, Takeuchi Y, Brinyiczki K, Zombori T, Oliva A, Fernandez-Ruiz A, Kozak G, Kincses ZT, Ivanyi B, Buzsaki G, Berenyi A. Direct effects of transcranial electric stimulation on brain circuits in rats and humans. Nat Commun. 2018 Feb 2;9(1):483. doi: 10.1038/s41467-018-02928-3. PMID 29396478
- [Background] Kim HC, Lee W, Kunes J, Yoon K, Lee JE, Foley L, Kowsari K, Yoo SS. Transcranial focused ultrasound modulates cortical and thalamic motor activity in awake sheep. Sci Rep. 2021 Sep 29;11(1):19274. doi: 10.1038/s41598-021-98920-x. PMID 34588588
- [Background] Feldman EL, Goutman SA, Petri S, Mazzini L, Savelieff MG, Shaw PJ, Sobue G. Amyotrophic lateral sclerosis. Lancet. 2022 Oct 15;400(10360):1363-1380. doi: 10.1016/S0140-6736(22)01272-7. Epub 2022 Sep 15. PMID 36116464

DOCUMENTS (1):
  • Study Protocol (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT06681610/Prot_000.pdf